CLINICAL TRIAL: NCT04942457
Title: Effects of Fasting in Fertility Treatment in Women
Brief Title: Feasibility and Safety of Fasting in Fertility Treatment
Acronym: KiWuA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Karl and Veronica Carstens Foundation (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KiWuA
Record Dates: First submitted 2021-05-10; First posted 2021-06-28 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Sub Fertility, Female; Fertility Disorders; Cycle Disorders Menstrual; Ovulation Disorder; Ovulation Absent; Ovulation Delayed; Ovulation; Failure or Lack of; Sub-fertility
Keywords: fasting; natural therapies; caloric restriction; lifestyle modification; dietary restriction; dietary intervention; prolonged fasting; weight loss; complementary medicine; integrative medicine
MeSH Terms: conditions — Infertility, Female; Menstruation Disturbances; Anovulation; Infertility; Fasting; Weight Loss | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: There are 2 parallel groups following different nutritional regimes. Additionally Qualitative Interviews with Patients and Doctors/Medical Staff.
Who Masked: Outcomes Assessor
Masking Description: It is not possible to mask a fasting intervention for the participant or the study personel. Therefore only outcome assessors are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (Experimental): Participants will be councelled and accompanied to follow a prolonged fasting regime of 7-10 days in an outpatient setting under medical supervision. Additionally qualitative interviews will be conducted by few participants in the experimental arm, as well as their respective Healthcare Providers (Doctors/Medical Staff).
  Interventions: Behavioral: Fasting
- Control group (No Intervention): waiting list, usual diet should be maintained

INTERVENTIONS:
Behavioral: Fasting — Prolonged fasting for 7-10 days (caloric intake <500 kcal in liquid form)
  Arms: Fasting

SUMMARY:
This exploratory study investigates fasting as a potential supportive therapy in infertility treatment for women suffering from infertility

DETAILED DESCRIPTION:
This 2-arm, randomized, controlled exploratory clinical trial aims to explore fasting as a novel supportive treatment in infertility. The participants will be randomized in two groups: fasting and waiting list. All groups will be trained and accompanied by medical experts and dieticians. In addition, qualitative interviews will be conducted including individual and focus group interviews with a subgroup of participants.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25 to 45 years
* Unfulfilled desire to have children >1 year
* declaration of consent
* 20 kg/m² ≤ BMI ≤ 40 kg/m²

Exclusion Criteria:

* Language barriers
* Previously known serious mental illness or cognitive impairment
* Patients with anatomical/organic damage and proven uterine abnormalities
* Eating disorders in the medical history
* Serious previous internal diseases
* Lack of internet access
* No consent to randomisation
* Participation in other studies

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — biological female sex
Enrollment: 34 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Qualitative interview analysis of fasting experience | in time frame of 24 weeks after fasting intervention
  individual and focus group interviews
pregancy rate | at baseline, after one month, at end of ovulation induction treatment (2-6 months) and 12 months after baseline
  pregnancy rate of the participants

SECONDARY OUTCOMES:
complication rates in pregnancy | 12 months after baseline
  complication rates monitored by the gynaecologist, if applicable
Hormonal status | at the beginning and end of each ovulatory cycle, for up to 12 months
  FSH, LH, Estrogen, Progesteron
HbA1c | baseline and at end of ovulation induction treatment (2-6 months), for up to 12 months
  serum parameter
WHO-5 | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  Quality of life
diet | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  questionnaire to examine dietary behaviour
mindfulness | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  MAAS-questionnaire, validated questionnaire to examine mindfulness
anxiety and depression | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  HADS-questionnaire, validated questionnaire to examine anxiety and depression
current mood | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  ASTS-questionnaire, validated questionnaire to examine current mood
experienced stress | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  Cohen-stress scale, validated questionnaire to examine experienced stress
physical fitness | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  questionnaire to examine physical fitness
quality of relationship | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  questionnaire to examine the relationship between the two partners desiring to have a child
psychological stress caused by the unfulfilled desire to have children | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  questionnaire to examine the psychological stress caused by the unfulfilled desire to have children
gratitude | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  validated questionnaire to examine gratitude
self-efficacy | at baseline, after fasting (1-3 weeks), after one month, at end of ovulation induction treatment (2-6 months)and 12 months after baseline
  ASKU, validated questionnaire to examine self-efficacy
abdominal ultrasound after liver wrap | before, during and after the fasting intervention
  sonography in a subgroup
rate of ovulations | at baseline, after one month, at end of ovulation induction treatment (2-6 months) and 12 months after baseline
  ovulation visible in sonography
liver function parameters | at baseline, after one month, at end of ovulation induction treatment (2-6 months), after 12 months
  serum liver enzymes
pyruvate in culture medium of oocytes, if applicable (in case of IVF/ICSI) | after in vitro fertilisation, if applicable during study period of one year
  chemical composition of culture medium (pyruvate)
glucose in culture medium of oocytes, if applicable (in case of IVF/ICSI) | after in vitro fertilisation, if applicable during study period of one year
  chemical composition of culture medium (glucose)
lactate in culture medium of oocytes, if applicable (in case of IVF/ICSI) | after in vitro fertilisation, if applicable during study period of one year
  chemical composition of culture medium (lactate)
Continuous Glucose Monitoring | 14 days after baseline
  Continuous Glucose Monitoring via CGM-Device in subgroup
Ketone bodies in breath | up to 4 days before, during and up to 7 days after fasting intervention
  Breath acetone, in subgroup
Cumulative drug dose for ovulation induction | baseline and until end of treatment for ovulation induction (2-6 months)
  Cumulative dosage of hormonal therapy for each assisted cycle of ovulation induction

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Hochschulambulanz für Naturheilkunde der Charité-Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: after the end of the study for 5 years
Access Criteria: on demand.